CLINICAL TRIAL: NCT00170079
Title: Prolonged Smoking Cessation Using Prescription Step Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert C. Klesges, Professor of Preventive Medicine, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1730-04; R01CA106667-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Step care vs. regular care (Experimental): Participants were randomized either to (1) Step care intervention, where smokers who failed to quit or who relapsed received increasingly intensive smoking cessation interventions; vs. (2) Regular care, where smokers who failed to quit or who relapsed received repeated intervention.
  Interventions: Behavioral: Smoking Cessation Intervention

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — A common approach to increasing long-term adherence and control of chronic medical problems such as hypertension in both general and preventive medicine is the concept of "step care." The purpose of this study is to evaluate the long-term efficacy of a step care model for smoking cessation that is disseminable in primary care settings. With that introduction, we propose the following specific aims:
  Aim 1: To enroll approximately 400 adult cigarette smokers recruited mainly from primary care settings;
  Aim 2: To randomize these participants to: 1) State of the Art Smoking Cessation + Recycling or 2) State of the Art Smoking Cessation + Step Care; and
  Aim 3: To evaluate the long-term (24 months post-randomization) relative success of the interventions. It is predicted that long-term cessation rates will be significantly higher in the step care condition.

SUMMARY:
Smoking is the number one preventable cause of morbidity and mortality in this nation. Unfortunately, more than 50% of those who quit following a smoking cessation intervention typically relapse within two weeks, with approximately 80% relapsing within six months. Therefore, tobacco use can be conceptualized as a chronic condition. As with many chronic medical problems, tobacco use interventions may benefit from a step care approach to treatment.

A total of 400 adult smokers will be enrolled in the study. Participants will be randomly assigned to one of two treatment conditions consisting of: 1) A State of the Art Smoking Cessation Intervention + Recycling or: 2) A State of the Art Smoking Cessation Intervention + Step Care. Long term smoking cessation will be assessed by self-report, exhaled carbon monoxide levels, and salivary cotinine. The primary endpoint of the study will be smoking abstinence rates at two-year follow-up. It is predicted that long-term cessation rates will be significantly higher in the step care condition than for those assigned to the recycling group.

DETAILED DESCRIPTION:
A common approach to increasing long-term adherence and control of chronic medical problems such as hypertension in both general and preventive medicine is the concept of step care. Despite a high degree of interest in applying the step care model to smoking cessation (Abrams et al., 1996; Hughes, 1994), little empirical work has been conducted utilizing this treatment approach. The purpose of this study is to evaluate the long-term efficacy of a step care model for smoking cessation that is disseminable in primary care settings. With that introduction, we propose the following specific aims:

Aim 1: To enroll approximately 400 adult cigarette smokers recruited mainly from primary care settings;

Aim 2: To randomize these participants to: 1) State of the Art Smoking Cessation + Recycling or 2) State of the Art Smoking Cessation + Step Care; and

Aim 3: To evaluate the long-term (24 months post-randomization) relative success of the interventions. It is predicted that long-term cessation rates will be significantly higher in the step care condition.

ELIGIBILITY:
Cigarette smokers who are 18 years of age or older, who self-report smoking at least 10 cigarettes each day, and who are willing to accept random assignment are eligible to participate. Potential participants must agree to commit to the study for at least 24 months, be screened and agree to potentially participate in more intensive interventions to help them stop smoking, and agree to not seek other treatment for smoking cessation during the treatment phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2005-04; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Long term smoking cessation using both prolonged and point prevalence abstinence criteria | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Klesges, Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Derived] Ebbert JO, Little MA, Klesges RC, Bursac Z, Johnson KC, Thomas F, Vander Weg MW. Step Care treatment for smoking cessation. Health Educ Res. 2017 Feb 1;32(1):1-11. doi: 10.1093/her/cyw051. PMID 28158558